CLINICAL TRIAL: NCT04256941
Title: INTERACT- Integrated Evaluation of Resistance and Actionability Using Circulating Tumor DNA in HR Positive Metastatic Breast Cancers
Brief Title: Aromatase Inhibitor Therapy With or Without Fulvestrant for the Treatment of HR Positive Metastatic Breast Cancer With an ERS1 Activating Mutation, the INTERACT Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Despite modifications, accrual was poor and the closed
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0287; NCI-2019-08825 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0287 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-01-21; First posted 2020-02-05 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Breast Carcinoma; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib; Anastrozole; Fulvestrant; Letrozole; palbociclib; ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (ribociclib, palbociclib, abemaciclib, fulvestrant) (Experimental): Patients receive ribociclib PO QD, palbociclib PO QD on days 1-21, and/or abemaciclib PO BID on days 1-28. Patients also receive fulvestrant IM for 2 injections over 1-2 minutes each on days 1 and 15 of cycle 1 and day 2 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Abemaciclib; Drug: Fulvestrant; Drug: Palbociclib; Drug: Ribociclib
- Arm II (ribociclib, palbociclib, abemaciclib, letrozole) (Active Comparator): Patients receive ribociclib orally PO QD, palbociclib PO QD on days 1-21, and/or abemaciclib PO BID on days 1-28. Patients also receive letrozole PO QD or anastrozole PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Abemaciclib; Drug: Anastrozole; Drug: Letrozole; Drug: Palbociclib; Drug: Ribociclib

INTERVENTIONS:
Drug: Abemaciclib — Given PO
  Other Names: LY-2835219; LY2835219; Verzenio
Drug: Anastrozole — Given PO
  Other Names: Anastrazole; Arimidex; ICI D1033; ICI-D1033; ZD-1033
  Arms: Arm II (ribociclib, palbociclib, abemaciclib, letrozole)
Drug: Fulvestrant — Given IM
  Other Names: Faslodex; Faslodex(ICI 182,780); ICI 182,780; ICI 182780; ZD9238
  Arms: Arm I (ribociclib, palbociclib, abemaciclib, fulvestrant)
Drug: Letrozole — Given PO
  Other Names: CGS 20267; Femara
  Arms: Arm II (ribociclib, palbociclib, abemaciclib, letrozole)
Drug: Palbociclib — Given PO
  Other Names: 6-Acetyl-8-cyclopentyl-5-methyl-2-((5-(piperazin-1-yl)pyridin-2-yl)amino)-8h-pyrido(2,3-d)pyrimidin-7-one; Ibrance; PD 0332991; PD 332991; PD 991; PD-0332991
Drug: Ribociclib — Given PO
  Other Names: Kisqali; LEE-011; LEE011

SUMMARY:
This phase II trial studies how well letrozole, anastrozole, or fulvestrant work when given together with ribociclib, palbociclib, and/or abemaciclib in treating patients with hormone receptor (HR) positive breast cancer that has spread to other places in the body (metastatic) and has an ERS1 activating mutation. Letrozole, anastrozole, ribociclib, palbociclib, and abemaciclib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Estrogen can cause the growth of breast cancer cells. Hormone therapy using fulvestrant may fight breast cancer by blocking the use of estrogen by the tumor cells. It is not yet known if giving letrozole, anastrozole, or fulvestrant with ribociclib, palbociclib, and/or abemaciclib will work better in treating patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess progression free survival (PFS) with transition to fulvestrant compared with continuing aromatase inhibitor (AI) therapy in patients with emergence of estrogen receptor 1 (ESR1) mutations in plasma.

SECONDARY OBJECTIVES:

I. To assess circulating tumor deoxyribonucleic acid (ctDNA) ESR1 mutant allele fraction (MAF) and kinetics with fulvestrant compared with AI.

II. To assess the prevalence of ESR1 mutations in patients with secondary resistance to endocrine therapy.

III. To correlate ctDNA with cancer antigens (CA) 15-3 tumor marker changes. IV. To assess overall survival (OS) with transition to fulvestrant compared with continuing AI therapy in patients with emergence of ESR1 mutations.

V. To assess PFS and time to next treatment (TTNT) on next line of therapy after progression on fulvestrant versus (vs.) AI in combination with CDKI.

EXPLORATORY OBJECTIVES:

I. Characterize other co-existing actionable genomic alterations of interest in relation to ESR1 and clinical outcomes.

II. To determine frequency of other actionable genomic alterations and frequency of enrollment on genotype-matched therapy.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive ribociclib orally (PO) once daily (QD), palbociclib PO QD on days 1-21, and/or abemaciclib PO twice daily (BID) on days 1-28. Patients also receive fulvestrant intramuscularly (IM) for 2 injections over 1-2 minutes each on days 1 and 15 of cycle 1 and day 2 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive ribociclib orally PO QD, palbociclib PO QD on days 1-21, and/or abemaciclib PO BID on days 1-28. Patients also receive letrozole PO QD or anastrozole PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelets >= 50 x 10^9/L
* Hemoglobin (Hb) >= 9 g/dL
* Total serum bilirubin =< 2.0 mg/dL
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x upper limit of normal (ULN) (=< 5 x ULN in patients with liver metastases)
* Serum creatinine =< 1.5 x ULN
* Activating ESR1 mutation (e.g. D538G, Y537S/N, S463P) identified on ctDNA. Novel ESR1 alterations allowed as per discretion of principal investigator (PI)
* On AI with CDK4/6 inhibitor (palbociclib, ribociclib, or abemaciclib) as first line therapy for metastatic breast cancer (MBC) for at least 12 months without evidence of clinical progression
* Patients with histologically confirmed HR positive (estrogen receptor [ER] positive [+] and/or progesterone receptor [PR]+ [> 10%]), MBC

Exclusion Criteria:

* Pregnant or lactating women
* Received prior therapy for MBC (except for AI use for up to 4 weeks prior to initiation of CDK4/6 inhibitor)
* Prior therapy with fulvestrant in the metastatic setting
* Corrected QT (QTc) interval > 480 msec, Brugada syndrome or known history of QTc prolongation or Torsade de Pointes
* Psychiatric illness which would limit informed consent
* Patients with de novo metastatic disease
* Patients who have any severe and/or uncontrolled medical conditions such as: unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction =< 6 months prior to enrollment, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease, active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, and active and chronic hepatitis (i.e. quantifiable hepatitis B virus [HBV]-DNA and/or positive hepatitis B surface antigen [HbsAg], quantifiable hepatitis C virus [HCV]-ribonucleic acid [RNA]), severe hepatic impairment (Child-Pugh C)
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy
* Expected survival < 6 months
* Any serious medical illness, other than that treated by this study, which would limit survival to less than 1 month
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study
* Patients who are currently part of or have participated in any clinical investigation with an investigational drug within 1 month prior to dosing
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, must use highly effective methods of contraception during the study and 8 weeks after the end of treatment. Highly effective contraception methods include combination of any two of the following: placement of an intrauterine device (IUD) or intrauterine system (IUS); barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository; total abstinence or; male/female sterilization
* Male patients whose sexual partner(s) are WOCBP who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senthilkumar Damodaran, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was opened to accrual on 5/31/2019. The study was intended for patients with ESR1 mutations. Despite modifications, accrual was poor and the closed to accrual on 8/24/2023
Pre-assignment Details: Of the 49 patients screened, 6 patients harbored ESR1 mutation. 4 patients were randomized to the study. 1 patient withdrew consent due to frequent travel/visits after randomization (AI arm). 1 patient was a screen fail due to elevated LFTs, and 1 patient passed away prior to study intervention)
Groups:
- Fulvestrant: Fulvestrant (Faslodex), a selective estrogen receptor antagonist, was initially indicated for treatment of HR positive MBC in post-menopausal women with disease progression following prior anti-estrogen therapy.
- Continuing AI After Randomization: CDK inhibitors e.g. palbociclib (Ibrance), ribociclib (Kisqali), and abemaciclib (verzenio) are approved for the first line treatment of HR positive advanced breast cancers in combination with aromatase inhibitors as well as in combination with fulvestrant with disease progression following prior endocrine therapy.
Period: Overall Study
Arm/Group | Fulvestrant | Continuing AI After Randomization
Started | 1 | 3
Completed | 0 | 0
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Death | 1 | 0
Not completed — Disease Progession | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fulvestrant | Continuing AI After Randomization | Total
Number analyzed (Participants) | 1 | 3 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 2 | 2
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 3 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Survival curves for PFS will be analyzed using the Kaplan-Meier method and survival difference across groups will be examined by log rank test. Will estimate the treatment comparison with 95% confidence intervals and p-value using Cox proportional hazards regression and we will assess the proportional hazard assumption using graphs of rescaled Schoenfeld residuals and related tests.
Time Frame: Up to 30 days
Population: No data was collected since despite modifications, accrual was poor and the closed. Outcome Measure has zero total analyzed at the protocol specified timepoint.
Arm/Group | Fulvestrant | Continuing AI After Randomization
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Circulating Tumor Deoxyribonucleic Acid (ctDNA) ESR1 Mutant Allele Fraction (MAF) and Kinetics
Description: Graphical analysis, such as scatter plots with Lowess smoothers, will be used to assess the correlative structure of outcomes and compare MAF between fulvestrant and aromatase inhibitor-treated groups. The Pearson correlation, or its non-parametric analogue, the Spearman correlation, will be used to estimate the linear correlation among variables.
Time Frame: Up to 30 days
Population: as for outcome 1
Arm/Group | Fulvestrant | Continuing AI After Randomization
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Prevalence of Emergence of Estrogen Receptor 1 (ESR1) Mutations
Description: Will be assessed by the secondary resistance of endocrine therapy.
Time Frame: Up to 30 days
Population: as for outcome 1
Arm/Group | Fulvestrant | Continuing AI After Randomization
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Changes in Cancer Antigens (CA) 15-3 Tumor Marker
Description: Will correlate ctDNA with CA 15-3 tumor marker changes.
Time Frame: Up to 30 days
Population: as for outcome 1
Arm/Group | Fulvestrant | Continuing AI After Randomization
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Overall Survival (OS)
Description: Survival curves for OS will be analyzed using the Kaplan-Meier method and survival difference across groups will be examined by log rank test. Will estimate the treatment comparison with 95% confidence intervals and p-value using Cox proportional hazards regression and we will assess the proportional hazard assumption using graphs of rescaled Schoenfeld residuals and related tests.
Time Frame: Up to 30 days
Population: as for outcome 1
Arm/Group | Fulvestrant | Continuing AI After Randomization
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Time to Next Treatment
Description: Will be assessed on next line of therapy after progression.
Time Frame: Up to 30 days
Population: as for outcome 1
Arm/Group | Fulvestrant | Continuing AI After Randomization
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 50 months and 3 weeks
Groups:
- Fulvestrant; Continuing AI After Randomization: CDK inhibitors e.g. palbociclib (Ibrance), ribociclib (Kisqali), and abemaciclib (verzenio) are approved for the first line treatment of HR positive advanced breast cancers in combination with aromatase inhibitors as well as in combination with fulvestrant with disease progression following prior endocrine therapy.
Arm/Group | Fulvestrant | Continuing AI After Randomization
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 1/1 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fulvestrant (N=1) | Continuing AI After Randomization (N=3)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Blurred Vision (General disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Cough (General disorders) | 1 | 0
Fall (Musculoskeletal and connective tissue disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1
ALT increased (Blood and lymphatic system disorders) | 0 | 2
Alkaline Phosphatase increased (Blood and lymphatic system disorders) | 0 | 1
Allergic Rhinitis (General disorders) | 0 | 1
AST increased (Blood and lymphatic system disorders) | 0 | 2
Hypercalcemia (Blood and lymphatic system disorders) | 0 | 1
Hyponatremia (Blood and lymphatic system disorders) | 1 | 1
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 | 2
White blood cell decreased (Blood and lymphatic system disorders) | 1 | 1
Vomiting (General disorders) | 1 | 0
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1 | 0
Creatinine increased (Blood and lymphatic system disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-08): https://cdn.clinicaltrials.gov/large-docs/41/NCT04256941/Prot_SAP_000.pdf